CLINICAL TRIAL: NCT01400893
Title: A Multi-Center, Randomized, Controlled, Pivotal Study To Assess the Safety and Efficacy of A Selective Cytopheretic Device (SCD) In Patients With Acute Kidney Injury (AKI)
Brief Title: Efficacy Study of a Selective Cytopheretic Device (SCD) in Patients With Acute Kidney Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: SeaStar Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCD-003
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Results first posted 2017-08-29 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Acute Kidney Injury
Keywords: Acute Renal Failure; Acute kidney injury; Acute tubular necrosis; Continuous Renal Replacement Therapy; Severe sepsis; Selective cytopheretic device
MeSH Terms: conditions — Acute Kidney Injury; Kidney Cortex Necrosis; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRRT + SCD (Experimental): Patients with a diagnosis of AKI requires CRRT will be randomized
  Interventions: Device: SCD
- CRRT alone (No Intervention): Patients with a diagnosis of AKI requires CRRT will be randomized

INTERVENTIONS:
Device: SCD — The selective cytopheretic device (SCD) is comprised of tubing, connectors and a hemofilter cartridge. The device is connected in series to a commercially available Continuous Renal Replacement Therapy (CRRT) device. Blood from the CRRT circuit is diverted after the CRRT hemofilter through to the extra capillary space (ECS) of the SCD. Blood circulates through this space and is returned to the patient via the venous return line of the CRRT circuit. Regional citrate anticoagulation is used for the entire CRRT and SCD blood circuits.
  Arms: CRRT + SCD

SUMMARY:
The purpose of this protocol is to evaluate the safety of a selective cytopheretic device (SCD) in patients that are on continuous renal replacement therapy (CRRT) for acute kidney injury (AKI).

DETAILED DESCRIPTION:
Acute kidney injury is a condition where the kidneys are not capable of producing adequate urine. Therefore, another way to remove waste from the body is needed to hopefully allow time for the kidneys to heal. One method of removing waste from the body is called Continuous Renal Replacement Therapy (CRRT) or variations of that therapy. This study will evaluate the safety of the device while it is connected to the CRRT tubing for up to 7 days. Patients will be followed up until day 60 following the treatment.

ELIGIBILITY:
Inclusion Criteria

1. A patient, or legal representative, has signed a written informed consent form.
2. Must be receiving medical care in an intensive care unit (e.g., ICU, MICU, SICU, CTICU, Trauma).
3. Age 18 to 80 years.
4. Females of child bearing potential who are not pregnant (confirmed by a negative serum pregnancy test) and not lactating if recently post-partum.
5. Must be receiving and tolerating CRRT therapy for a minimum of 4 hours, but not longer than 24.
6. Expected to remain in the ICU for at least 96 hours after evaluation for enrollment.
7. A clinical diagnosis of ATN due to hemodynamic or toxic etiologies. ATN is defined as Acute Kidney Injury occurring in a setting of acute ischemic or nephrotoxic injury with oliguria (average <20 mL/hr) for >6-12 hours or: an increase in serum creatinine ≥2 mg/dL (≥1.5 mg/dL in females) over a period of ≤4 days. (Note: Prerenal, hepatorenal, vascular, interstitial, glomerular, and obstructive etiologies are excluded on clinical or other diagnostic grounds.)
8. Presence of at least one non-renal organ failure or present sepsis as defined in Appendix C.
9. All patients must be able to tolerate regional citrate anticoagulation.

Exclusion Criteria:

1. Irreversible brain damage based on available historical and clinical information.
2. Presence of any organ transplant at any time.
3. Acute or chronic use of circulatory support device such as LVADs, RVADs, BIVADs, ECMO.
4. Presence of preexisting advanced chronic renal failure (i.e., ESRD) requiring chronic renal replacement therapy prior to this episode of acute kidney injury.
5. AKI occurring in the setting of burns, obstructive uropathy, allergic interstitial nephritis, acute or rapidly progressive glomerulonephritis, vasculitis, hemolytic-uremic syndrome, thrombotic thrombocytopenic purpura (TTP), malignant hypertension, scleroderma renal crisis, atheroembolism, functional or surgical nephrectomy, hepatorenal syndrome, cyclosporine or tacrolimus nephrotoxicity.
6. Metastatic malignancy which is actively being treated or may be treated by chemotherapy or radiation during the subsequent three month period after study therapy.
7. Chronic immunosuppression (e.g., HIV/AIDS, chronic glucocorticoid therapy >20 mg/day prednisone equivalent on a chronic basis). The acute use of glucocorticoids is permissible.
8. Severe liver failure as documented by a Child-Pugh Liver Failure Score >12 (see Appendix F).
9. Currently in Do Not Resuscitate (DNR) status or DNR status anticipated within the next 7 days.
10. Currently in Comfort measures Only or Comfort Measures Only status anticipated within next 7 days.
11. Patient is moribund or chronically debilitated for whom full supportive care is not indicated.
12. Patient not expected to survive 28 days because of an irreversible medical condition. (This is not restrictive to AKI, and may include situations such as the presence of irreversible brain damage, untreatable malignancy, inoperable life threatening condition, or any condition to which therapy is regarded as futile by the PI.)
13. Any medical condition that the Investigator thinks may interfere with the study objectives.
14. Physician refusal.
15. Patient is a prisoner.
16. Dry weight of >150 kg.
17. More than one hemodialysis treatment during this hospital admission or prior to transfer from an outside hospital.
18. Platelet count <30,000/mm3 at time of screening.
19. Concurrent enrollment in another interventional clinical trial. Patients enrolled in clinical trials where only measurements and/or samples are taken (NO TEST DEVICE OR TEST DRUG USED) are allowed to participate.
20. Use of any other Investigational drug or device within the previous 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - University of Alabama Birmingham, Birmingham, Alabama
  - UCLA, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of Florida, Gainesville, Florida
  - University of Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Mississippi, Jackson, Mississippi
  - Washington University, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - Mount Sinai School of Medicine, New York, New York
  - Sanford Health, Fargo, North Dakota
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University Of South Carolina, Charleston, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - Erlanger Hospital, Chattanooga, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - University of Texas, Houston, Texas
  - INOVA Health Care Services, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Result] Tumlin JA, Galphin CM, Tolwani AJ, Chan MR, Vijayan A, Finkel K, Szamosfalvi B, Dev D, DaSilva JR, Astor BC, Yevzlin AS, Humes HD; SCD Investigator Group. A Multi-Center, Randomized, Controlled, Pivotal Study to Assess the Safety and Efficacy of a Selective Cytopheretic Device in Patients with Acute Kidney Injury. PLoS One. 2015 Aug 5;10(8):e0132482. doi: 10.1371/journal.pone.0132482. eCollection 2015. PMID 26244978
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4526678/

RESULTS

PARTICIPANT FLOW:
Groups:
- CRRT + SCD: Patients with a diagnosis acute kidney injury with multiorgan failure requiring CRRT will be randomized
  SCD: The selective cytopheretic device (SCD) is comprised of tubing, connectors and a hemofilter cartridge. The device is connected in series to a commercially available Continuous Renal Replacement Therapy (CRRT) device. Blood from the CRRT circuit is diverted after the CRRT hemofilter through to the extra capillary space (ECS) of the SCD. Blood circulates through this space and is returned to the patient via the venous return line of the CRRT circuit. Regional citrate anticoagulation is used for the entire CRRT and SCD blood circuits.
- CRRT Alone: Patients with a diagnosis of acute kidney injury and multiorgan failure requiring CRRT will be randomized
Period: Overall Study
Arm/Group | CRRT + SCD | CRRT Alone
Started | 69 | 65
Completed | 42 | 38
Not Completed | 27 | 27
Not completed — Death | 27 | 21
Not completed — Lost to Follow-up | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- CRRT + SCD: Patients with a diagnosis acute kidney injury with multiorgan failure requiring CRRT will be randomized.
  SCD: The selective cytopheretic device (SCD) is comprised of tubing, connectors and a hemofilter cartridge. The device is connected in series to a commercially available Continuous Renal Replacement Therapy (CRRT) device. Blood from the CRRT circuit is diverted after the CRRT hemofilter through to the extra capillary space (ECS) of the SCD. Blood circulates through this space and is returned to the patient via the venous return line of the CRRT circuit. Regional citrate anticoagulation is used for the entire CRRT and SCD blood circuits.
- CRRT Alone: Patients with a diagnosis acute kidney injury with multiorgan failure requiring CRRT will be randomized.
- Total: Total of all reporting groups
Arm/Group | CRRT + SCD | CRRT Alone | Total
Number analyzed (Participants) | 69 | 65 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (13.1) | 53.5 (14.7) | 55.4 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 42 | 40 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 14 | 29
  White | 53 | 48 | 101
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 69 | 65 | 134

OUTCOME MEASURES:

1. Primary Outcome: The Primary Clinical Efficacy Endpoint in This Trial is All Cause Mortality Through 60 Days Post-randomization.
Description: All cause mortality through day 60 post-randomization.
  The outcome data reported here describe the mortality at Day 60 (primary endpoint) of the treated subjects which received the recommended ionized calcium (riCa) for ≥ 90% of treatment time.
Time Frame: Day 60 following treatment initiation
Population: Outcome data is reported for those subjects in which the calcium levels were maintained in the protocol's recommended range (≤0.4 mmol/L) for greater or equal to 90% of the therapy time.
Measure: Count of Participants; unit: Participants
Arm/Group | CRRT + SCD | CRRT Alone
Number analyzed (Participants) | 19 | 27
Participants
  Alive | 16 | 16
  Dead | 3 | 11

2. Secondary Outcome: Renal Replacement Therapy Dependency at Day 60.
Description: RRT dependency at day 60 is defined as patient not receiving any form of intermittent or continuous renal replacement therapy at 60 days post enrollment in the study with no plans for additional intermittent or continuous renal replacement therapy.
Time Frame: Day 60 following treatment initiation
Population: per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- CRRT + SCD: Patients with a diagnosis of AKI will be randomized
  SCD: The selective cytopheretic device (SCD) is comprised of tubing, connectors and a hemofilter cartridge. The device is connected in series to a commercially available Continuous Renal Replacement Therapy (CRRT) device. Blood from the CRRT circuit is diverted after the CRRT hemofilter through to the extra capillary space (ECS) of the SCD. Blood circulates through this space and is returned to the patient via the venous return line of the CRRT circuit. Regional citrate anticoagulation is used for the entire CRRT and SCD blood circuits.
- CRRT Alone: Patients with a diagnosis of AKI will be randomized
Arm/Group | CRRT + SCD | CRRT Alone
Number analyzed (Participants) | 19 | 26
Participants | 3 | 15

ADVERSE EVENTS:
Time Frame: Up to 7 days of SCD treatment or control. This time frame differs from the primary outcome measure of 60 day mortality since therapy was provided up to 7 days of SCD treatment. The adverse events were captured only during SCD treatment times since device related events would occur at that time frame. ITT patients are included in this table.
Description: Trial results showed that a number of enrollees in the treated and control arms deviated from protocol requiring regional citrate anticoagulation due to a national shortage of injectable CaCl2. The Primary Outcome is reported for patients who were treated per protocol.
  Two subjects enrolled to CRRT alone arm were not treated, so not counted in SAEs. 60 Day Mortality does not include 6 subjects LTFU.
  Other Adverse Events were not collected.
Arm/Group | CRRT + SCD | CRRT Alone
All-Cause Mortality (participants affected / at risk) | 27/69 | 21/59
Serious Adverse Events (participants affected / at risk) | 45/69 | 40/63
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRRT + SCD (N=69) | CRRT Alone (N=63)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 8 (8) | 3 (3)
Cardiac disorders (Cardiac disorders) | 12 (12) | 10 (10)
Gastrointestinal disorders (Gastrointestinal disorders) | 4 (4) | 6 (6)
General disorders and administration site conditions (General disorders) | 4 (4) | 7 (7)
Infections and infestations (Infections and infestations) | 12 (12) | 10 (10)
Injury, poisoning and procedural conplications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Investigations (Investigations) | 0 (0) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1) | 3 (3)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (10)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Vascular disorders (Vascular disorders) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes